CLINICAL TRIAL: NCT05407389
Title: An Open-Label Rollover Extension Phase 2 Clinical Trial To Evaluate The Long-Term Safety And Efficacy Of KT-301 (Formerly US-APR2020) In Subjects With CKD IV Completing The US-APR2020-01 Study
Brief Title: Rollover Extension Clinical Trial To Evaluate The Long-Term Safety And Efficacy Of KT-301 (Formerly US-APR2020) In Subjects With CKD IV Completing The US-APR2020-01 Study
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Logistics, company reorganization.
Sponsor: Kibow Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: US-APR2020-02
Record Dates: First submitted 2022-05-27; First posted 2022-06-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Disease stage4

STUDY DESIGN:
Intervention Model Description: This is an extension open-label multicenter study to evaluate the long-term safety and efficacy of KT-301 (formerly US-APR2020) in patients with CKD Stage IV. KT-301 will be administered orally at 2 capsules per day (a total dose of 90 Billion CFUs per day of the Live BioTherapeutic).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KT-301 (formerly US-APR2020) (Experimental)
  Interventions: Drug: KT-301 (formerly US-APR2020)

INTERVENTIONS:
Drug: KT-301 (formerly US-APR2020) — KT-301 (formerly US-APR2020) will be administered orally at 2 capsules per day (a total dose of 90 Billion CFUs per day of the Live BioTherapeutic).

SUMMARY:
This is an Open-Label Rollover Extension Clinical Trial to Evaluate the Long-Term Safety and Efficacy of KT-301 (formerly US-APR2020) in Subjects With CKD IV Who Completed the US-APR2020-01 Study

DETAILED DESCRIPTION:
Kidney diseases are a global public health problem that affects over 200 million people worldwide. It is estimated that about 30 million adults in the United States have Chronic Kidney Disease (CKD) and most are undiagnosed. In addition, CKD represents the ninth leading cause of death in the United States. Kidney diseases also represent great socioeconomical cost worldwide. In the United States, treating Medicare beneficiaries with CKD costed over $79 billion, and treating people with End Stage Kidney Disease (ESKD) costed an additional $35 billion in 2016. To date, there is no cure for CKD.

CKD is accompanied by altered pathogenic gut bacteria, inflammation, and accumulation of uremic toxins in the blood. These blood uremic toxins can diffuse passively into the bowel. Scientific research has shown that probiotic bacteria could metabolize various uremic toxins such as urea, uric acid and creatinine. In addition, by supplementing the gut microbiome with probiotic bacteria, it is possible to metabolize the nitrogenous waste products and other toxins which diffuse into the gut, and thus lower levels of inflammation and blood uremic toxins.

KT-301 (formerly US-APR2020) is a probiotic formulation of bacteria intended to restore the gut bacteria balance to improve the removal of uremic toxins in the bowel in CKD patients.

This is an open label, multicenter, rollover extension study to provide KT-301 to subjects who were previously enrolled into and completed the placebo-controlled study, US-APR2020-01. Subjects will roll over to the long-term extension study at the last visit of the US-APR-2020-01 study. All subjects who completed the US-APR2020-01 study will be eligible to enroll in this study.

The purpose of this open-label study is to evaluate the long-term safety and efficacy of the live biotherapeutic product, KT-301, in the management of patients with CKD Stage IV.

ELIGIBILITY:
Inclusion Criteria:

* Completion of US-APR2020-01 study
* Adults between the ages of 18-80 years

Exclusion Criteria:

* Did not participate in the placebo-controlled study US-APR2020-01
* Withdrew from US-APR2020-01 study prior to completing the 6 months treatment for any reason
* Unwilling or unable to visit the site for the follow-up visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the long-term safety of KT-301 (formerly US-APR2020) in patients with Chronic Kidney Disease (CKD) Stage IV | 6 months
  Presence of adverse events in less than 10% of the study population, as a measure of safety Chronic Kidney Disease (CKD) Stage IV
Evaluate the clinical efficacy of KT-301 (formerly US-APR2020) in patients with Chronic Kidney Disease (CKD) Stage IV | 6 months
  Arresting the decline of eGFR as per NKF-USFDA guidelines following date of roll- over transition until study competition, compared to baseline (End of study for US- APR2020-01) as a measure of clinical efficacy

SECONDARY OUTCOMES:
Evaluate changes in basic blood uremic metabolic markers | 6 months
Evaluate changes in complete blood count and hematology parameters | 6 months
Reduction in C-Reactive Protein (CRP) levels following date of roll-over transition until study competition | 6 months
Percent change in rating scale (Modified SF36 QOL questionnaire) from roll-over transition until study competition (at 24-weeks) | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Jadedstone Clinical Research, Silver Spring, Maryland
  - Kidney Michigan, Saginaw, Michigan
  - South Carolina Clinical Research, Orangeburg, South Carolina
  - Almeda Medical Clinic, Houston, Texas
  - Mendez Center for Clinical Research, Woodbridge, Virginia